CLINICAL TRIAL: NCT00031564
Title: Phase II Study of a B7-1 Gene-Modified Autologous Tumor Cell Vaccine and Systemic IL-2 for Patients With Stage IV Renal Cell Carcinoma
Brief Title: Phase II Study of a B7-1 Gene-Modified Autologous Tumor Cell Vaccine and Systemic IL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12207; NCI-5090 (Other: NCI); NCI-G00-1872 (Other: NCI); 0001386 (Other: OBA)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Cancer
Keywords: stage IV; renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interleukin-2; aldesleukin; B7-1 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine Therapy With Interleukin-2 (Experimental): At approximately 3-6 weeks after surgery, patients receive B7-1 gene-modified autologous tumor cell vaccine subcutaneously (SC) once on days 1, 29, and 57. At 6 weeks after the first vaccination, patients receive interleukin-2 (IL-2) SC five days a week for 6 weeks (days 43-82). Patients with stable or responding disease after day 106 may receive additional vaccinations in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Interleukin-2; Biological: B7-1

INTERVENTIONS:
Biological: Interleukin-2
  Other Names: Aldesleukin; IL-2
Biological: B7-1
  Other Names: gene-modified autologous tumor cell vaccine

SUMMARY:
RATIONALE: Vaccines made by inserting a laboratory-treated gene into a person's tumor cells may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining vaccine therapy with interleukin-2 may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining vaccine therapy with interleukin-2 in treating patients who have stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the percentage of patients with stage IV renal cell carcinoma with a reduction in tumor size after treatment with B7-1 gene-modified autologous tumor cell vaccine and interleukin-2.
* Determine the immunogenicity of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the local and systemic toxicity of this regimen in these patients.

OUTLINE: Tumor tissue for vaccine preparation is obtained when patients undergo palliative surgical resection of primary tumor or therapeutic resection of metastasis.

At approximately 3-6 weeks after surgery, patients receive B7-1 gene-modified autologous tumor cell vaccine subcutaneously (SC) once on days 1, 29, and 57. At 6 weeks after the first vaccination, patients receive interleukin-2 (IL-2) SC five days a week for 6 weeks (days 43-82). Patients with stable or responding disease after day 106 may receive additional vaccinations in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 weeks after the last dose of IL-2.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV renal cell carcinoma

  * Symptomatic primary tumor or resectable metastasis
* Measurable disease post resection
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL
* Hematocrit greater than 30%

Hepatic:

* Bilirubin less than 2 times normal
* SGOT less than 3 times normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No evidence of active myocardial ischemia, prior myocardial infarction, or arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindications to surgical resection
* No history of immunodeficiency disease
* No known allergy to penicillin

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior interleukin-2, interferon alfa, or other biologic agent allowed

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent corticosteroids (except for replacement doses for adrenal insufficiency)

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No concurrent immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2000-05; Primary Completion 2005-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Who Have a Reduction in the Size of Their Measurable Metastatic Tumors | 4 years
  The primary objective of this phase II trial involving 30 patients will be to determine tumor response rates. The immunogenicity of the treatment will be assessed by ELISPOT assays performed on the patients' peripheral blood lymphocytes, and by an immunohistochemical analysis of DTH skin tests site biopsies performed 48 hours after the intradermal injection of autologous, unmodified tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Scott J. Antonia, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Fishman M, Hunter TB, Soliman H, Thompson P, Dunn M, Smilee R, Farmelo MJ, Noyes DR, Mahany JJ, Lee JH, Cantor A, Messina J, Seigne J, Pow-Sang J, Janssen W, Antonia SJ. Phase II trial of B7-1 (CD-86) transduced, cultured autologous tumor cell vaccine plus subcutaneous interleukin-2 for treatment of stage IV renal cell carcinoma. J Immunother. 2008 Jan;31(1):72-80. doi: 10.1097/CJI.0b013e31815ba792. PMID 18157014